CLINICAL TRIAL: NCT00396617
Title: Voice Prosthesis Made in Porous Titanium After Total Laryngectomy or Pharyngolaryngectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: OseoAnvar (Unknown); Réseau National des Technologies de Santé (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3736
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Pharyngeal Neoplasms; Laryngeal Neoplasms; Carcinoma
Keywords: Laryngeal or pharyngo-laryngeal's carcinoma,; voice prosthesis tracheooesophageal shunt,; titanium beads,; cellular colonization; Laryngeal or pharyngo-laryngeal's carcinoma
MeSH Terms: conditions — Pharyngeal Neoplasms; Laryngeal Neoplasms; Carcinoma; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: prothesis voice — The device may be used for patient using another type of voice prosthesis, of for patient undergoing total laryngectomy. This device is definitively placed in two parts:The first one is introduced in the puncture (TEP) through the esophagus (retrograde way). The second part is then clipped on the first one through the tracheotomy orifice (anterograde way).A third part containing the valve can then be clipped in the prosthesis and easily removed in order to change it as often as necessary.
Procedure: total laryngectomy — The second part is then clipped on the first one through the tracheotomy orifice (anterograde way).A third part containing the valve can then be clipped in the prosthesis and easily removed in order to change it as often as necessary.

SUMMARY:
The benefits of this new material, as demonstrated in animal studies and preliminary studies in man, could provide the answer to problems encountered by surgeons in the field of phonatory implants. This novel application is a step towards resolving the very real problems which still exist in the field today. The functional concept, which will allow better control over integrating implants in tissue, should also, it is hoped, favour cellular colonization, thereby fulfilling a currently unmet medical need. The aim is to avoid well-identified potential complications linked to the use of silicone-only implants (with or without a surface coating), like leakage around the prosthesis (by cellular colonization), and so reduce the risk of protrusion/extrusion of the prosthesis as far as possible, and to avoid trauma to the peri-prosthetic tissues by repeated interventions

ELIGIBILITY:
Inclusion criteria:

* age more than 18
* total laryngectomy or pharyngo-larynctomy

Exclusion criteria:

* pregnant women-age less than 18
* major pulmonary bronchitis
* major neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2007-12; Primary Completion 2013-09 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Clinical measures concerning peri and intra prosthetic leakage | days 8,15,21,30 - months : 2 ,4,6,8, 10, 12, 15,18,21,24,30, 36

SECONDARY OUTCOMES:
Phonology's measures | months 1, 3,12

CONTACTS AND LOCATIONS:
Overall Officials: Christian DEBRY, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg, France